CLINICAL TRIAL: NCT00157053
Title: Evaluation of Pharmacokinetics, Safety, Efficacy and Immunogenicity of rAHF-PFM in Previously Treated Hemophilia A Patients - A Continuation Study
Brief Title: Study of Pharmacokinetics, Efficacy and Safety of a Recombinant and Protein-Free Factor VIII (rAHF-PFM) in Hemophilia A Patients - A Continuation of Clinical Study 069901
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060102
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hemophilia A
Keywords: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

INTERVENTIONS:
Drug: Antihemophilic factor, recombinant, manufactured protein-free

SUMMARY:
The purpose of this study is to evaluate whether rAHF-PFM is safe and effective in the treatment of hemophilia A subjects. The study consists of 2 parts: Part 1 is a pharmacokinetic and safety study, and Part 2 is an evaluation of efficacy and safety. The study is open to patients who completed Baxter Study 069901.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed Baxter protocol 069901
* Subject is HIV-1 seronegative or, if HIV-1 seropositive, has a CD4+ lymphocyte count >= 400/mm3 documented within three months of the screening visit
* Subject (and his legally acceptable representative, in the case of study participants >= 10 and < 18 years of age) has been informed of the nature of the study, agreed to its provisions, and signed and dated the informed consent form approved by the appropriate IRB/IEC and Baxter

Exclusion Criteria:

* The subject received factor VIII products other than rAHF-PFM upon completion of Baxter protocol 069901
* The subject developed an inhibitor to factor VIII, measured in the central laboratory, during Baxter protocol 069901. An inhibitor is defined as a Bethesda titer > 1.0 or, if Bethesda titer < 1.0, confirmation using the Nijmegen modification of the Bethesda assay with a titer > 0.6
* The subject is scheduled to receive an immunomodulating drug other than anti-retroviral chemotherapy (e.g., a-interferon, steroids) during the course of the study
* The subject is identified by the investigator as being unable or unwilling to cooperate with study procedures

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2001-11-22 (Actual); Primary Completion 2004-08-03 (Actual); Study Completion 2004-08-03 (Actual)

PRIMARY OUTCOMES:
Terminal phase half-life for Recombinant Antihemophilic Factor (rAHF-PFM) | Within 30 minutes prior to the pharmacokinetic infusion and at 1 hour ± 5 minutes, 9 ± 1 hour, 24 ± 2 hours, and 48 ± 2 hours after the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (24):
- United States (11):
  - Mountain States Regional Hemophilia and Thrombosis Center, Aurora, Colorado
  - Childrens Healthcare of Atlanta Blood Bank, Atlanta, Georgia
  - Comprehensive Bleeding Disorders Center, Peoria, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Michigan State University, East Lansing, Michigan
  - University of Medicine & Dentistry of New Jersey, New Brunswick, New Jersey
  - Cornell Medical Center, New York, New York
  - Mt. Sinai Medical School, New York, New York
  - Children's Hospital Medical Center Pharmacy, Cincinnati, Ohio
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Puget Sound Blood Center, Seattle, Washington
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- KU Leuven Universitaire Ziekenhuizen, Leuven, Belgium
- University of Alberta, Calgary, Alberta, Canada
- Hôpital Edouard Herriot, Lyon, France
- Germany (3):
  - Klinikum der J. W. Goethe - Universität, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Innenstadt der Universität München, Munich
- Ospedale Maggiore di Milano, Milan, Italy
- University Hospital MAS, Malmo, Sweden
- United Kingdom (4):
  - The Royal Free Hospital, London, England
  - Central Manchester Healthcare NHS Trust, Manchester, England
  - The Churchill Hospital, Oxford, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Shapiro A, Gruppo R, Pabinger I, Collins PW, Hay CR, Schroth P, Casey K, Patrone L, Ehrlich H, Ewenstein BM. Integrated analysis of safety and efficacy of a plasma- and albumin-free recombinant factor VIII (rAHF-PFM) from six clinical studies in patients with hemophilia A. Expert Opin Biol Ther. 2009 Mar;9(3):273-83. doi: 10.1517/14712590902729392. PMID 19216617